CLINICAL TRIAL: NCT02797782
Title: Study of the Long Term Efficacy of Recombinant Hepatitis B Vaccine in Young Adults 20-22 Years After the Primary Vaccination in Nile Delta of Egypt
Brief Title: Study of the Long Term Efficacy of Recombinant Hepatitis B Vaccine in Nile Delta of Egypt
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Consultant liver and GIT diseases- Tanta university hospital, Tanta University
Organization: Tanta University (Other)
Other Study IDs: HBV vaccine
Record Dates: First submitted 2016-06-08; First posted 2016-06-13 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Hepatitis B Vaccines
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Detection of anti HBs antibody titer — All samples will be analyzed for anti HBs antibody titer using ELISA kits.

SUMMARY:
More than two billion individuals have serological evidence of hepatitis B virus (HBV) infection worldwide. Of these, 240 million are chronic carriers and approximately 786,000 hepatitis B related deaths occur annually.

Currently available hepatitis B vaccines are extremely safe and have an efficacy of >90 percent against all HBV serotypes and genotypes. Thus, HBV infection can potentially be eradicated through global vaccination. A positive immune response to the vaccine is defined as the development of hepatitis B surface antibody (anti-HBs) at a titer of >10 mIU/mL.

Although anti-HBs titers decrease with time, the duration of protection is long. Protection has been estimated to persist for up to 22 years after the primary vaccination schedule. Protection from clinical disease, despite declining or even undetectable anti-HBs levels, is probably due to the priming of memory cells, which are capable of eliciting an anamnestic response when challenged. This is supported by the rapid increases in anti-HBs titers in previously vaccinated individuals who administered booster injections.

DETAILED DESCRIPTION:
A significant proportion of the vaccinated population loses both the protective levels of anti-HBs and an anamnestic response. Recommendations for booster vaccination have been proposed in a European consensus statement. Countries like the Netherlands, Germany, Spain, France and Belgium recommend a booster dose depending on the post-vaccination anti-HBs titer. In the UK, a single booster dose is recommended five years after primary vaccination.

In Egypt, the routine infant immunization for hepatitis B virus started in 1992, and was given at 2nd, 4th and 6th months of age. In the present study the investigators will investigate the long term efficacy of hepatitis B vaccination in young adults 20 to 22 years after the primary vaccination in Nile Delta of Egypt.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-22 years
* Administration of HBV vaccine during routine infant immunization (2nd, 4th, 6th months after birth)

Exclusion Criteria:

* Overt co-morbid condition
* Treatment with immune-modulatory or immune-suppressive drugs

Ages: 20 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Age 20-22 years
  * Administration of HBV vaccine during routine infant immunization (2nd, 4th, 6th months after birth)
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-12 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Number of individuals with protective anti-HBs antibody titers | 1 year
  Number of individuals having protective anti-HBs antibody titers

CONTACTS AND LOCATIONS:
Overall Officials: Asem Elfert, Prof, Principal Investigator — Hepatology and gastroenterology dept.-Tanta; Reham Elkhouly, Consultant, Study Chair — Division of Gastroenterology and Hepatology- Tanta; Rehab Badawi, Consultant, Study Chair — Hepatology and gastroenterology dept.-Tanta; Walaa Elkhalawany, Consultant, Study Chair — Hepatology and gastroenterology dept.-Tanta; Mona Watany, Consultant, Study Chair — clinical pathology dept.-Tanta; Sherief Abd-Elsalam, Consultant, Study Chair — Hepatology and gastroenterology dept.-Tanta
Locations (1):
- Sherief Abd-Elsalam, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided